CLINICAL TRIAL: NCT02180269
Title: A Double-Blind, Placebo-Controlled, Randomized, Single-Ascending Dose Study to Investigate the Safety, Tolerability and Pharmacokinetics of JNJ-54861911 in Healthy Japanese Male Subjects
Brief Title: A Safety, Tolerability and Pharmacokinetics Study of JNJ-54861911 in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR104614; 54861911ALZ1006 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2014-07-01; First posted 2014-07-02 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
Keywords: Healthy; JNJ-54861911; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Experimental): Single oral dose of either JNJ-54861911, 25 milligram (mg) tablet or matched placebo tablet on Day 1.
  Interventions: Drug: JNJ-54861911 (25 mg); Drug: Placebo
- Cohort B (Experimental): Single oral dose of either JNJ-54861911, 50 mg (2*25 mg tablets) or matched placebo tablets on Day 1.
  Interventions: Drug: JNJ-54861911 (50 mg); Drug: Placebo
- Cohort C (Experimental): Single oral dose of either JNJ-54861911, 100 mg (4*25 mg tablets) or matched placebo tablets on Day 1.
  Interventions: Drug: JNJ-54861911 (100 mg); Drug: Placebo

INTERVENTIONS:
Drug: JNJ-54861911 (25 mg) — Single oral dose of JNJ-54861911, 25 mg on Day 1.
  Arms: Cohort A
Drug: JNJ-54861911 (50 mg) — Single oral dose of JNJ-54861911, 50 mg on Day 1.
  Arms: Cohort B
Drug: JNJ-54861911 (100 mg) — Single oral dose of JNJ-54861911, 100 mg on Day 1.
  Arms: Cohort C
Drug: Placebo — Single oral dose of placebo matched to JNJ-54861911 on Day 1.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK, study of the way a drug enters and leaves the blood and tissues over time) of single-ascending oral doses of JNJ-54861911 in healthy Japanese male participants.

DETAILED DESCRIPTION:
This is a single-center, randomized (study medication assigned to participants by chance), double-blind (neither Investigator nor participant knows which treatment the participant receives), placebo controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), study of a single-ascending dose of JNJ-54861911 in participants between 55 to 75 years of age. The duration of study will be approximately 2 to 6 weeks per participant. The study consists of 3 periods: Screening period (28 to 2 days prior to dose administration); Double-blind Treatment period (participants will receive either a single oral dose of JNJ-54861911 or placebo as tablets under fasted conditions); and a Follow-up visit period (7 to 14 days after dose administration). All the eligible participants will be assigned to any of following 3 cohorts: Cohort A (single oral dose of JNJ-54861911, 25 milligram [mg] or placebo); Cohort B (single oral dose of JNJ-54861911, 50 mg or placebo); Cohort C (single oral dose of JNJ-54861911, 100 mg or placebo). Each cohort will include 8 participants. Participants in each cohort will be randomly assigned to receive either a single oral dose of JNJ-54861911 (n = 6) or placebo (n = 2). Blood samples will be collected pre-dose and over 96 hours (that is up to Day 5) after dosing for understanding the PK characteristics of JNJ-54861911. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed an informed consent document indicating they understand the purpose of and procedures required for the study, and are willing to participate in the study
* A man, who is sexually active with a woman of child-bearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator, and must not donate sperm during the study and for 90 days after receiving the study drug
* Body mass index between 18 and 30 kilogram (kg) per square meter
* Blood pressure (supine for 5 minutes) between 90 and 150 millimeter of mercury (mm Hg) systolic, and no higher than 90 mm Hg diastolic
* Must be healthy on the basis of physical and neurological examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening or admission (up to Day 1 predose)

Exclusion Criteria:

* History of or current liver or renal impairment, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, dermatological (at the puncture site) or metabolic disturbances
* History of spontaneous, prolonged and severe bleeding of unclear origin
* History of epilepsy or fits
* History of human immunodeficiency virus (HIV) antigen/antibody positive, or tests positive for HIV at screening

Ages: 55 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs) | Screening up to 14 days after last dose administration or early withdrawal
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 14 days after last dose administration, that were absent before treatment or that worsened relative to pretreatment state.
Maximum Plasma Concentration (Cmax) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-administration of drug on Day 1
  The Cmax is the maximum observed plasma concentration.
Time to Reach Maximum Concentration (Tmax) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-administration of drug on Day 1
  The Tmax is time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-administration of drug on Day 1
  The AUC (0-last) is area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (Clast).
Apparent Clearance (CL/F) | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-administration of drug on Day 1
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.

SECONDARY OUTCOMES:
Cerebrospinal Fluid (CSF) Amyloid-Beta Concentration | 24 hours pre-administration of drug on Day -1, 24 hours post-administration of drug on Day 2
  Amyloid-beta (biomarker, supposed to be a key feature in the pathogenesis of Alzheimer's disease) levels in CSF will be explored.
Plasma Amyloid-Beta Concentration | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 hours post-administration of drug on Day 1
  Amyloid-beta (biomarker, supposed to be a key feature in the pathogenesis of Alzheimer's disease) levels in plasma will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Fukuoka, Japan